CLINICAL TRIAL: NCT03502408
Title: Perfusion Imaging Evaluation for Ischemic Stroke on 6-24 Hours Undergoing Endovascular Thrombectomy
Acronym: PESET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: yan2017-150
Record Dates: First submitted 2018-03-29; First posted 2018-04-18 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Stroke, Acute Cerebral Infarction
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Endovascular Thrombectomy (Experimental): Procedure: Endovascular Thrombectomy Device: Trepo trevor Retriever Device: Solitaire™ FR Revascularization Device
  Interventions: Procedure: Endovascular Thrombectomy

INTERVENTIONS:
Procedure: Endovascular Thrombectomy — Procedure: Endovascular Thrombectomy Device: Trepo trevor Retriever Device: Solitaire™ FR Revascularization Device
Procedure: Endovascular Thrombectomy — Procedure:Endovascular Thrombectomy Device: Solitaire™ FR Revascularization Device

SUMMARY:
This study aims to evaluate the hypothesis that thrombectomy devices plus medical management leads to superior clinical outcomes in acute ischemic stroke patients at 90 days as compared to medical management alone in appropriately selected subjects with the Target Mismatch Profile and an MCA (M1 and M2 segment) or ICA occlusion or BA who have endovascular thrombectomy initiated between 6-24 hours after last seen well.

DETAILED DESCRIPTION:
Study design is a prospective, single-center study of acute ischemic stroke patients with large artery occlusion in 6-24 hours of stroke onset. According to patients or their family members' willing, patients who meet the inclusion criteria will be assigned to endovascular thrombectomy group with approved devices (only the devices listed in this protocol are approved for us) plus standard medical therapy or control group (standard medical therapy alone) after undergoing either CT Perfusion or MR Perfusion studies. Patients who have evidence of an ICA or MCA M1 or M2 or BA occlusion and a Target Mismatch Profile will be enrolled.

The intent of this study is to support thrombectomy beyond the currently labeled 8 hour indicated time limit in wake up, unclear onset, and late presenting ischemic stroke subjects, who currently have no other option besides medical management of their symptoms, with careful selection.

The study will enroll up to 55 patients. The primary endpoint, the modified Rankin Score, will be assessed at 3 months.

ELIGIBILITY:
Inclusion Criteria:

Clinical Inclusion Criteria:

1. Clinical signs and symptoms consistent with the diagnosis of an acute ischemic stroke
2. Age ≥18 years
3. NIHSS ≥ 6
4. Endovascular thrombectomy can be initiated (femoral puncture) between 6 and 24 hours after time last know well
5. No significant pre-stroke disability (pre-stroke mRS must be ≤ 3 )
6. Patient/Legally Authorized Representative has signed the Informed Consent form

Imaging Inclusion Criteria:

1. ICA or MCA-M1 or MCA-M2 or BA occlusion (carotid occlusions can be cervical or intracranial with or without tandem MCA lesions) as evidenced by MRA or 4D-CTA
2. Target Mismatch Profile on CT perfusion or MR perfusion: ischemic core volume is ≤ 70 ml, mismatch ratio is >/= 1.2 )

Exclusion Criteria:

Clinical Exclusion Criteria:

1. Other serious, advanced, or terminal illness (investigator judgment) or life expectancy is less than 90 days
2. Subject with a co-morbid disease or condition that would confound the neurological and functional evaluations or compromise survival or ability to complete follow-up assessments
3. Unable to undergo a contrast brain perfusion scan with either MRI or CT
4. Pregnant
5. Known serious sensitivity to radiographic contrast agents
6. Treated with rtPA >6 hours after time last known well
7. Known hereditary or acquired hemorrhagic diathesis, coagulation factor deficiency; recent oral anticoagulant therapy with INR > 3 (recent use of one of the new oral anticoagulants is not an exclusion if estimated GFR > 30 ml/min).
8. Seizures at stroke onset if it precludes obtaining an accurate baseline NIHSS
9. Current participation in another investigational drug or device treatment study
10. Known hereditary or acquired hemorrhagic diathesis, coagulation factor deficiency
11. Any other condition that, in the opinion of the investigator, precludes an endovascular procedure or poses a significant hazard to the subject if an endovascular procedure was performed.

Neuroimaging Exclusion Criteria:

1. ASPECTS score <6 on non-contrast CT (if patient is enrolled based on CT perfusion criteria)
2. Evidence of intracranial tumor (except small meningioma), acute intracranial hemorrhage, neoplasm, subarachnoid hemorrhage, or arteriovenous malformation
3. Significant mass effect with midline shift
4. Evidence of internal carotid artery dissection
5. Intracranial stent implanted in the same vascular territory, known history of arterial tortuosity, and/or other arterial disease that precludes the safe deployment/removal of the thrombectomy device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Good Functional Independence | 90 days
  This outcome will look at the proportion of patients with mRS 0-2 at day 90.

SECONDARY OUTCOMES:
Death | 90 days
  Death
Symptomatic Intracranial Hemorrhage | 24 hours
  Defined as NIHSS worsening of 4 or more points associated with ICH within 24 hours of randomization

CONTACTS AND LOCATIONS:
Overall Officials: MIN LOU, Ph.D., Study Director — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No